CLINICAL TRIAL: NCT03339765
Title: Piloting a Serious Game to Improve Self-Advocacy Among Women With Advanced Cancer
Brief Title: Self-Advocacy Serious Game in Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Teresa Thomas, PhD, RN, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO17070414
Record Dates: First submitted 2017-11-03; First posted 2017-11-13 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Cancer Stage III; Ovarian Cancer Stage IV; Breast Cancer Stage IV; Cervical Cancer Stage IIIB; Cervical Cancer Stage IVA; Cervical Cancer Stage IVB; Endometrial Cancer Stage III; Endometrial Cancer Stage IV; Vulvar Cancer, Stage III; Vulvar Cancer, Stage IV; Vaginal Cancer Stage III; Vaginal Cancer Stage IVA; Vaginal Cancer Stage IVB
Keywords: Self-advocacy; Advanced cancer; Serious games; Self-management
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious game intervention (Experimental): Participants randomized to the intervention will receive the Strong Together serious game program on a tablet computer. The goal of this serious game is to teach the participant how to advocate for her needs relate to her cancer and treatment. The research team will send participants weekly notifications for 12 weeks to alert them that a new serious game session is available and encourage them to complete one session per week.
  Interventions: Behavioral: Strong Together serious game
- Enhanced care as usual (No Intervention): If randomized to the enhanced care as usual arm, the research team will give participants a paper-based self-advocacy patient brochure published by the National Coalition for Cancer Survivorship. This guide is not a part of usual care, but is freely available on the Internet.

INTERVENTIONS:
Behavioral: Strong Together serious game — The Strong Together serious game program is an interactive, immersive education program in which participants quickly learn the behaviors of self-advocacy and the potential consequences of self-advocating or not. Participants will receive weekly game sessions to play at home for three months.
  Arms: Serious game intervention

SUMMARY:
Self-advocacy, defined as the ability of a patient to get her needs and priorities met in the face of a challenge, is an essential skill but not all women with advanced cancer are able to do it. We want to instruct women with advanced cancer who have low self-advocacy to self-advocate for their health and well-being. We will test a new "serious game" or video program that teaches self-advocacy skills through interactive, situation-based activities. The goal of the Strong Together serious game is to engage participants in challenges commonly experienced by women with advanced cancer, offer them choices to self-advocate or not, and directly show them the health and social benefits of self-advocating and the negative consequences of not self-advocating. Through engaging in the Strong Together program, participants vicariously learn the essential skills of self-advocacy, understand the downstream effects of using or not using these skills, and learn distinct behaviors that they can then use to address their own challenges.

DETAILED DESCRIPTION:
Background: When faced with the challenges of advanced cancer, women must advocate (or stand up) for their needs and priorities. However, there are no interventions to promote self-advocacy among female patients with advanced cancer. Preliminary work has developed a theoretically-based, psychometrically-strong measure of self-advocacy (the Female Self-Advocacy in Cancer Survivorship (FSACS) Scale) and demonstrated correlations with symptom burden and healthcare utilization. Serious games offer a novel mechanism by which to deliver interactive, engaging health education that links users' choices to consequences so that users learn a desired skill. The fully-automated Strong Together self-advocacy serious game may allow women with advanced cancer to learn self-advocacy skills and therefore improve their health outcomes.

Objective/Hypothesis: The purpose of this pilot randomized controlled trial (RCT) is to evaluate the feasibility, acceptably, and preliminary efficacy of the Strong Together serious game.

Specific Aims:

Specific Aim 1: To evaluate the feasibility and acceptability of the 3-month Strong Together intervention.

* Benchmark 1: At least 75% of participants will engage in at least 8 out of the 12 serious game sessions.
* Benchmark 2: At least 80% of participants will find the intervention acceptable based on ratings of perceived satisfaction and ease of use, as well as feedback from qualitative exit interviews.

Specific Aim 2: To explore the differences in self-advocacy and symptom burden between groups over time.

• Research Question: Do patients who receive the intervention report improved self-advocacy and lower symptom burden compared to those assigned to enhanced care as usual?

Study Design: This pilot RCT will recruit (N=84) women from cancer clinics at the University of Pittsburgh Medical Center. Eligibility criteria include: female; age ≥ 18 years; diagnosis of Stage III or IV gynecological or Stage IV breast cancer within the past 3 months; 6-month prognosis; Eastern Cooperative Oncology Group score of 0-1; and ability to read and write in English. Measures will be collected at baseline, 3 months, and 6 months. Randomization (2:1) will occur to the 3-month Strong Together intervention group or the enhanced care as usual group. Feasibility will be assessed by calculating percentages of the intervention's dosage, engagement, recruitment, retention, and data completion. Acceptability will be assessed through exit interviews and an acceptability scale. Preliminary efficacy will be measured by exploring differences in self-advocacy and symptom burden scores and calculating point and interval estimates between the groups at 3 and 6 months.

Cancer Relevance: This study represents a unique opportunity to address the lack of self-advocacy interventions, reduce the risks of women with low self-advocacy, and guide an adequately-powered RCT to educate women with advanced cancer to self-advocate.

ELIGIBILITY:
Inclusion Criteria:

* Female

  -≥18 years
* Diagnosed with Stage III or IV gynecological or Stage IV breast cancer within the past 3 months being treated with non-curative intent
* Have at least a 6-month life expectancy (as determined by their oncologist)
* Eastern Cooperative Oncology Group performance score of 0 to 2 (per health record or oncologist)
* Able to read and write in English

Exclusion Criteria:

* On hospice at the time of recruitment
* Impaired cognition (per health record)
* Other active, unstable mental health disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion criteria are based on cancer diagnoses which primarily occur in women (gynecological and breast cancer).
Enrollment: 78 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Number of participants who engage in at least 8 out of the 12 serious game sessions | 3 months
  We will calculate the number of participants in the intervention group who complete two-thirds (66.7%) of the intervention sessions as a measure of intervention feasibility. We will accept that we achieved adequate feasibility if at least 75% of participants engage in at least eight out of the twelve serious game sessions.
Number of participants who find the intervention acceptable based on ratings of the Post Study System Usability Questionnaire and qualitative interviews. | 3 months
  We will accept that we achieved adequate acceptability if at least 80% of participants find the intervention acceptable based on the Post Study System Usability Questionnaire scores and if no issues are raised during the qualitative interviews and feedback that cannot be revised prior to the future trial.

SECONDARY OUTCOMES:
Change in patient self-advocacy as assessed by the Female Self-Advocacy in Cancer Survivorship Scale. | Baseline, 3 months, and 6 months
  We anticipate that self-advocacy scores will increase (improve) among participants in the intervention group compared to the enhanced care as usual group.
Change in symptom burden as assessed by the MD Anderson Symptom Inventory scale. | Baseline, 3 months, and 6 months
  We anticipate that symptom burden scores will decrease (improve) among participants in the intervention group compared to the enhanced care as usual group.
Change in healthcare utilization as assessed by participants' number of hospital admissions, emergency room visits, and primary care visits in the past three months. | Baseline, 3 months, and 6 months
  We anticipate that the frequency of healthcare utilization will decrease (improve) among participants in the intervention group compared to the enhanced care as usual group.
Change in quality of life as assessed by the Functional Assessment of Cancer Therapy-General scale. | Baseline, 3 months, and 6 months
  We anticipate that quality of life will increase (improve) among participants in the intervention group compared to the enhanced care as usual group.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa H Thomas, PhD, RN, Principal Investigator — University of Pittsburgh School of Nursing
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No